CLINICAL TRIAL: NCT00514566
Title: Is Polydioxanone 'THE' Suture of Choice for Midline Abdominal Closure? Results of a Prospective Randomized Clinical Trial
Brief Title: PDS vs Polyamide for Midline Abdominal Closure
Acronym: PPMAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unacceptable incidence of wound dehiscence in the PDS group
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChristianMCLudhiana
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Laparotomy
Keywords: Polyamide; Polydioxanone; Midline; Abdominal; Closure
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Surgical Patient undergoing midline laparotomy closure
  Interventions: Device: Suture for midline abdominal closure

INTERVENTIONS:
Device: Suture for midline abdominal closure — closure with Polyamide or Polydioxanone
  Other Names: Ethicon Inc., Loop no. 1, 150 cm suture length

SUMMARY:
Within the last decade the customary trend of using non absorbable sutures has changed, with numerous studies and meta-analyses advocating the use of slowly absorbable sutures, claiming comparable wound strength with significantly lower incidence of wound complications. It was the objective of this randomized clinical trial to compare two universally accepted suture materials, the non-absorbable Nylon and the slowly absorbable Polydioxanone for midline abdominal closure in the Indian context.

DETAILED DESCRIPTION:
64 patients undergoing midline laparotomy were allocated, using block randomization, to mass closure of the abdominal wall with continuous polyamide (34 patients) or continuous polydioxanone (30 patients).

There was an alarmingly higher incidence of wound dehiscence in the PDS group requiring secondary suturing (Nylon 0; PDS 5). Mid-way through the trial, an interim analysis was performed which revealed an unacceptably high incidence of wound dehiscence in the PDS group. This necessitated a premature curtailment of the study. There was, however, a statistically significantly higher incidence of scar pain in the Nylon group (Nylon 9; PDS 1).

There is a need for a study with larger series, and PDS as a choice of suture for midline wound closure cannot be recommended.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 12 years of age undergoing midline abdominal fascial closure using a continuous technique in the Department of Surgery, Christian Medical College and Hospital

Exclusion Criteria:

* All patients under 12 years of age
* Gynaecological operations
* Abdominal wall hernia repair

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Wound Complications associated with suture material used for closure- Wound Dehiscence, Wound Infection, Incisional Hernia, Suture Sinus, Scar Pain | 2 years

SECONDARY OUTCOMES:
Factors independent of suture materials responsible for wound complications such as age, gender, type of surgery, degree of contamination, surgeon, and presence of a stoma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Kapoor, MS(Gen Surg), Study Chair — Christian Medical College and Hospital, Ludhiana, India
Locations (1):
- Christian Medical College and Hospital, Ludhiana, Punjab, India